CLINICAL TRIAL: NCT06701279
Title: Role of Electrocardiogram Abnormalities in Prediction of Mortality in Patients with Isolated Traumatic Brain Injury
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yomna Mohamed Abdellatif, resident doctor at Emergency medicine unit Faculty of Medicine, Assiut University, Assiut University
Other Study IDs: ECG Traumatic brain Injury
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Traumatic Brain Injury
Keywords: Electrocardiogram
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- group 1: Patients with brain traumatic injury

SUMMARY:
Most common causes of ECG changes, from surgical view, are extradural haemorrhage , intracerebral haemorrhage, intraventricular haemorrhage and subarachnoid haemorrhage. A previous study reprorted ST-T wave changes in 41.5% of acute brain injury patients. In another paper , the prolonged QT interval was existed in (42.4%) of the included patients, ST depression (3.4%), ST elevation (3.4%),and morphologic end-repolarization abnormalities (10.2%). One paper reported that inverted T Wave was prevalent in 2% of the study population on admission and 0 after 24 hours of admission. The prognostic value of ECG abnormalities on the TBI patient fate is still under research.

In this study we aim to observe any correlation between ECG changes in patients with isolated TBI who will attend to ED in Assiut university hospital.

Aim of study:

Predictive value in mortality of ECG abnormalities in patients with isolated Traumatic brain injury (TBI).

DETAILED DESCRIPTION:
Traumatic brain Injury (TBI) is a brain affection occurring due to whether external blunt or penetrating trauma applied to the head. It may results from gun-shot, car accident, falling, assault or even suicide. Recently, TBI is considered one of the major leading causes to disability and death . Also variant neurological diseases e.g. neurodegenerative and demential diseases are reported as long term complication of TBI . According to Global Burden of Diseases (GBD) TBI is defined as an external force applied to the head that causes varying degrees of damage to the brain and classified into mild, moderate and sever types according to Glasgow Coma Score (GCS). Globally in 2014, epidemiological estimations reported 2.53 million TBI-related emergency department (ED) visits from CDC documentation and in 2019, incidence of TBI was 27.16 million accounting for 346 per 100,000 populations and affecting the global economy what made it a major public health problem.

As TBI is a comorbid, disabling and a significant factor in world-wide morality; a lot of research papers are conducted concerning pathophysiology, epidemiology, risk factors, management, and treatment especially in neurosurgical field. From etiological view, falling is the most common factor for TBI followed by motor and motor-cyclic accidents. Concerning of age, the most vularnable group is elderly people who aged above 65 years followed by pediatrics aged below 4 years .

Epidemiologic estimates about TBI and its mortality rate faces difficulty because of some mild cases don't go to ED and some of sever cases died after accident.

in the last decade, research papers reported electrocardiogram (ECG) changes and abnormalities in patients with brain injury whether it is pathological as stroke or traumatic by external force. The cause of ECG changes in TBI patients is still searched but one of the explanations suggesting that it occurs due to autonomic instability and cardiac dysfunction as myocardial ischemic - like changes.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥ 18 years.
* In-patient diagnosed with any degree of isolated TBI.

Exclusion Criteria:

* Pediatric TBI patients aged below 18 years.

  * Poly-traumatic patients.
  * Cardiac arrest after trauma before arrival ED .
  * Cardiac patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with brain traumatic injury who will match the eligible criteria will be included. In this study, patients with trauma who will attend to emergency department will be subjected to primary and secondary survey. On attendance, after primary survey completion; ECG will be conducted to all patients. Any patients will have cardiac tamponade, aortic injury or for cardio-thoracic emergent operation will be excluded. Also, pediatric patients aged below 18 years old or adults get arrested before ED arrival will be excluded.
Sampling Method: Probability Sample
Enrollment: 54 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Mortality rate of TBI patients with ECG changes | 48 hours
  Number of deaths' among TBI patients with ECG changes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beverland DE, Rutherford WH. An assessment of the validity of the injury severity score when applied to gunshot wounds. Injury. 1983 Jul;15(1):19-22. doi: 10.1016/0020-1383(83)90156-0. PMID 6885141
- [Background] GBD 2019 Mental Disorders Collaborators. Global, regional, and national burden of 12 mental disorders in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet Psychiatry. 2022 Feb;9(2):137-150. doi: 10.1016/S2215-0366(21)00395-3. Epub 2022 Jan 10. PMID 35026139
- [Background] Gu D, Ou S, Liu G. Traumatic Brain Injury and Risk of Dementia and Alzheimer's Disease: A Systematic Review and Meta-Analysis. Neuroepidemiology. 2022;56(1):4-16. doi: 10.1159/000520966. Epub 2021 Nov 24. PMID 34818648